CLINICAL TRIAL: NCT05442671
Title: Home Exercise Training in Pediatric Pulmonary Hypertension
Brief Title: iTONE Trial (exercIse Training in pulmONary hypertEnsion) Exercise Program for Pediatric PH
Acronym: iTONE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-018168; 1K23HL150337-01A1 (NIH)
Record Dates: First submitted 2022-06-24; First posted 2022-07-05 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary Hypertension
Keywords: Actigraphy
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home exercise intervention (Other): * Personalized 16 week home exercise program - aerobic exercise for 20 minutes per day/4 days per week and light resistance exercise using resistance bands 3 days per week.
  * Aerobic sessions will include walking, biking, or light jogging, depending on access to facilities/equipment and weather.
  * Smartwatch for the length of the intervention and a heart rate monitor during exercise sessions.
  * Max heart rate prescribed will be 80% of that on recent cardiopulmonary exercise test (at most 150 beats/min).
  * Heart rate monitor will sync with the smartwatch.
  * Activity and heart rate data will be transmitted to the study team via a data hub connected to the participant's home internet modem several times per week.
  * Periodic text messaging to remind participants to wear the watch, sync the data, or adhere to heart rate goals, to ask about symptoms, or to support activity progress.
  * Multiple ways to contact the study team with questions or concerns.
  Interventions: Behavioral: Exercise intervention

INTERVENTIONS:
Behavioral: Exercise intervention — 16-week home exercise intervention, enriched by mobile health technology

SUMMARY:
Children with pulmonary hypertension (PH) engage in less physical activity than their peers. This is a concern since adult data support exercise as a non-pharmacologic treatment for PH. Despite adult data, therapeutic exercise has not been widely adopted in pediatric PH. Investigators have previously demonstrated that children with PH have less skeletal muscle mass in association with worse exercise performance. Interventions to increase physical activity and skeletal muscle mass may improve exercise performance and quality of life in children with PH. This study will use wearable activity monitoring devices to promote physical activity in a 16-week pilot intervention in children and teenager with PH.

DETAILED DESCRIPTION:
Pediatric pulmonary hypertension (PH) is a rare disease, affecting 2-16 per million children. Without treatment, pulmonary vascular disease leads to right ventricular cardiac failure and death. Survival has improved with pharmacologic advances, however, 5-year survival from diagnosis is still only about 75%. Even with increased survival, pediatric PH is a severe, chronic illness with physical and psychosocial burdens affecting the quality of life of children and families. Exercise intolerance is nearly universal and adversely affects quality of life. While exercise physiology is complex, skeletal muscle deficits and dysfunction are important factors associated with exercise intolerance in adults with PH. The contraction of the skeletal muscle pump helps increase pulmonary blood flow at the initiation of upright exercise in the normal circulation. Low skeletal muscle mass and muscle dysfunction may impair this mechanism in PH. Investigators previously demonstrated low skeletal muscle mass in association with worse exercise performance in children with PH and identified this as an intervention target. As children with PH engage in less moderate and vigorous physical activity compared to healthy peers, we hypothesize that increasing physical activity could increase skeletal muscle mass and lead to improved exercise performance.

Recent trials have demonstrated improved exercise performance and functional class in adults with PH undertaking prescribed exercise training. Pediatric data are limited to a single, small study in which exercise performance improved after a 16-week home exercise program. That intervention did not include skeletal muscle assessment, wearable activity monitors, or specified behavioral theory, as does the current proposal. The characteristics of the optimal PH exercise program are not clear as prior studies often failed to provide sufficient detail to enable reproducibility. Most programs have been hospital-based, some with additional at-home components. Duration has varied from 4-15 weeks. Programs have included aerobic, resistance, and respiratory exercise. Patient adherence has been inconsistently assessed. While wearable activity monitors have been used to assess activities of daily living of PH patients, they have not been employed in PH exercise programs. In youth, practical concerns of developmental differences, access to facilities or equipment, and parental time commitment must be considered, and home programs may be critical to avoiding missed school and work.

Newer technologic advances enable remote monitoring of physical activity in the home setting. Wearable accelerometer sensors with wireless transmission capabilities allow us to measure relevant endpoints from a patient's daily life. In this study, participants will undergo baseline assessment of muscle mass and strength and quality of life prior to a 16-week home exercise program, enriched by mobile health technology. Investigators will use a wrist-worn accelerometer paired with periodic text messages to measure activity, obtain daily downloads, and engage patients to promote adherence. Assessment of muscle mass and strength and quality of life will be repeated after the intervention. This real-time monitoring of adherence and feedback to the patient represent fundamental changes in PH treatment paradigms that can significantly enhance efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-18 years
* PH World Health Organization (WHO) diagnostic groups 1, 2, 3, or 4 (pulmonary arterial hypertension, PH due to left heart disease, PH due to lung disease, chronic thromboembolic PH)
* WHO functional class I or II
* Ambulatory status
* Mean pulmonary to systemic arterial pressure ratio <0.75 on most recent cardiac catheterization
* Stable PH medication regimen for 3 months prior to the intervention
* Home Wifi connection
* Mobile device in family capable of receiving text messages

Exclusion Criteria:

* WHO functional class III or IV
* Single ventricle physiology
* Moderate to severe renal disease (>stage 3)
* Severe hepatic impairment [aspartate aminotransferase (AST)/alanine transaminase (ALT) > 2x upper limit of normal]
* Current pregnancy
* Significant developmental delay/inability to comply with verbal instructions to complete the study procedures

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in moderate to vigorous physical activity (MVPA) | Pre-exercise intervention and Post intervention (within 2 weeks of completion of the 16-week exercise intervention)
  Change in MVPA (min/day) will be measured by smartwatch accelerometer from baseline over the course of the intervention

SECONDARY OUTCOMES:
Change in leg lean mass Z-score (LLMZ) | Pre-exercise intervention and Post intervention (within 2 weeks of completion of the 16-week exercise intervention)
  LLMZ will be measured by densitometry. LLMZ is a percentile score with scores -2 to 2 considered typical
Change in muscle strength | Pre-exercise intervention and Post intervention (within 2 weeks of completion of the 16-week exercise intervention)
  Upper extremity strength will be measured by handgrip dynamometer. Lower extremity strength will be measured by Biodex across the knee and ankle
Change in quality of life score | Pre-exercise intervention and Post intervention (within 2 weeks of completion of the 16-week exercise intervention)
  Score measured by completion of PedsQL questionnaire. Scores range from 0-100 with higher scores indicating better quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No